CLINICAL TRIAL: NCT07394907
Title: The Effectiveness of Gamified Metaverse-Based Training on Patient Safety for Nursing Students: A Mixed Methods Study
Brief Title: The Effectiveness of Gamified Metaverse-Based Training on Patient Safety for Nursing Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, BETUL SAHIN KILINC, lecturer, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 17162298600-374
Record Dates: First submitted 2026-01-31; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Gamification; Nursing Education; Patient Safety; Mixed Method Implementation Study

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gamified metaverse-based educational application (Experimental)
  Interventions: Behavioral: Gamified metaverse-based educational application
- Traditional-based education practice (No Intervention)

INTERVENTIONS:
Behavioral: Gamified metaverse-based educational application — Students in the intervention group will receive gamified metaverse-based training.
  Arms: Gamified metaverse-based educational application

SUMMARY:
Introduction: Patient safety issues, such as medication errors, healthcare-associated infections, unsafe surgical procedures, and diagnostic errors, can negatively impact the quality of healthcare and patient outcomes due to preventable risks. There is a need for innovative, interactive educational approaches to ensure the lasting acquisition of patient safety competencies in nursing students and to strengthen their transfer to the clinical environment. Aim: This study aims to evaluate the effect of gamified metaverse-based training on patient safety competencies in nursing students and to assess student opinions regarding metaverse-based training. Method: The research will be conducted using a mixed-methods design. The quantitative phase will be an experimental design including intervention and control groups, pre-test-post-test, and a one-month follow-up (retention test). The research will be conducted between February 2026 and May 2026 with second-year students studying in the Spring semester of 2025-2026 at Başkent University Nursing Department in Ankara. According to G*Power calculations, a minimum sample size of 52 was found; considering a possible 10% loss, the total sample size was planned as 60 students (intervention=30, control=30). All participants will take the Patient Safety Knowledge Level Test (pre-test) and the Patient Safety Competency Self-Assessment Tool before the training. This will be followed by 2 hours of traditional theoretical training on patient safety; the intervention group will also receive gamified metaverse-based training via Spatial.io for two weeks. Post-tests will be administered after the training and one month later. Data collection tools include the Demographic Information Form, the Patient Safety Knowledge Level Test, the Patient Safety Competency Self-Assessment Tool (PSCS), and focus group interviews to be conducted in the intervention group. Quantitative data will be analyzed through within-group and between-group comparisons; qualitative data will be analyzed using thematic analysis, and the findings will be interpreted holistically. Findings (Expected): Gamified metaverse-based training is expected to provide a greater increase in mean scores on the Patient Safety Knowledge Level Test (PSL) and total and sub-dimension scores (knowledge-skills-attitudes) of nursing students compared to the control group, and to support the retention of these results.

Conclusion: This study is expected to generate evidence regarding the effectiveness of gamified metaverse-based training in improving patient safety competencies in nursing education and to contribute to the structuring of patient safety training in a more integrated, student-centered, and sustainable manner.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agreeing to participate in the research,
* Being a second-year undergraduate nursing student,
* Being able to understand and speak Turkish,
* Having healthy hearing, vision, and speech.

Exclusion Criteria:

* The student voluntarily wishing to withdraw from the study
* The student ceasing to use the metaverse space during the study period
* Filling out the survey form incompletely.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
The Patient Safety Knowledge Level Test | Before the intervention, within 1 hour after the intervention, and one month after the intervention.
  The Patient Safety Knowledge Level Test, developed by Buldak and Tüzer (2025), will be administered as follows: a pre-test to determine students' current knowledge level regarding patient safety, a post-test (1) within one hour following the metaverse application, and a 1st retention test/post-test-2 one month later to measure the retention of learning. The Patient Safety Knowledge Level Test consists of 20 multiple-choice questions with 5 options each, related to patient safety knowledge. A minimum score of 0 and a maximum score of 100 are possible on this test. A higher score indicates an increased knowledge level.
Patient Safety Competency Self-Evaluation Tool | Before the intervention, within 1 hour after the intervention, and one month after the intervention.
  The scale was developed to measure nursing students' knowledge, skills, and attitudes regarding patient safety through self-assessment, and its Turkish adaptation was done by Eskici et al. (2021). The multidimensional scale consists of 3 dimensions (Knowledge=6 items, Skills=21 items, Attitudes=14 items), 12 factors, and a total of 41 items; items are scored on a 5-point Likert scale according to the dimensions (Knowledge: 1=I have no knowledge-5=I know very well; Skills: 1=I cannot do it at all-5=I can do it very easily; Attitudes: 1=I strongly disagree-5=I strongly agree). Items 38 and 39 are reverse-scored, and evaluation is done based on total and sub-dimension/factor average scores due to the multidimensional nature of the scale; higher scores indicate better patient safety competence. The internal consistency of the Turkish form was found to be high (total Cronbach's alpha=0.941; sub-dimensions 0.642-0.932).

SECONDARY OUTCOMES:
Focus Group Interview Questions (interview) | within 1 week after the intervention
  Focus group interview questions, formulated by researchers based on the literature (Gülcan, 2021; Jeon et al., 2020; Verkuly et al., 2020) to collect qualitative data, will be used for data collected using the focus group interview technique. This form will be finalized after necessary adjustments are made based on expert opinions.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Ankara, Turkey (Türkiye)